CLINICAL TRIAL: NCT02255110
Title: A Phase II, Single-arm, Japanese Multicenter Trial of TH-302 in Combination With Doxorubicin in Subjects With Locally Advanced Unresectable or Metastatic Soft Tissue Sarcoma
Brief Title: A Japanese Trial of TH-302 in Subjects With Locally Advanced Unresectable or Metastatic Soft Tissue Sarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision due to negative result of Phase 3 study TH-CR-406/SARC021
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Threshold Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR200592-008
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-07

CONDITIONS: Soft Tissue Sarcoma
Keywords: Locally Advanced Unresectable or Metastatic Soft Tissue Sarcoma; TH-302; Doxorubicin; Evofosfamide
MeSH Terms: conditions — Sarcoma | interventions — TH 302; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TH-302 and doxorubicin (Experimental)
  Interventions: Drug: TH-302; Drug: Doxorubicin

INTERVENTIONS:
Drug: TH-302 — TH-302 will be administered at a dose of 300 milligram per square meter (mg/m^2) by intravenous infusion over 30 minutes on Days 1 and 8 of every 21-day cycle until the evidence of significant treatment-related toxicity or progressive disease.
Drug: Doxorubicin — Doxorubicin will be administered at a dose of 75 mg/m^2 by intravenous injection (over at least 5 minutes) or by intravenous infusion over 6-96 hours on Day 1 of every 21-day cycle starting 2 to 4 hours after completion of TH-302 administration until the evidence of significant treatment-related toxicity or progressive disease.

SUMMARY:
This is a Phase 2, single-arm, Japanese multicenter trial to evaluate the safety, tolerability, and efficacy of TH-302 in combination with doxorubicin in subjects with locally advanced unresectable or metastatic soft tissue sarcoma (STS).

ELIGIBILITY:
Inclusion Criteria:

* Male or female Japanese subjects greater than or equal to (>=) 15 years of age
* Able to understand the purposes and risks of the trial and has signed or, if appropriate, the subject's parent or legal guardian has signed a written informed consent form approved by the Institutional Review Board (IRB) or Independent Ethics Committee (IEC)
* Pathologically confirmed diagnosis of STS of the histopathologic types as specified in the protocol
* Locally advanced unresectable or metastatic disease with no standard curative therapy available and for whom treatment with single agent doxorubicin is considered appropriate
* Recovered from reversible toxicities of prior therapy
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (at least one target lesion outside of previous radiation fields or progressed within a previous radiation field)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of at least 3 months
* Acceptable liver function, renal function, hematologic status (without growth factor support for neutropenia or transfusion dependency), and cardiac function as specified in the protocol
* All women of childbearing potential must have a negative serum pregnancy test and all subjects must agree to use effective means of contraception (surgical sterilization or the use of barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an intrauterine device, intrauterine device [IUD]) with their partner from entry into the trial through 6 months after the last dose. Post-menopausal women must meet the criteria of 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum follicle-stimulating hormone (FSH) levels greater than (>) 35 international units per liter (IU/L)

Exclusion Criteria:

* Low grade tumors according to standard grading systems (for example, American Joint Committee on Cancer [AJCC] Grade 1 and 2 or Fédération Nationale des Centres de Lutte Contre le Cancer [FNCLCC] Grade 1)
* Prior systemic therapy for advanced or metastatic STS (neoadjuvant therapy followed by surgical resection and adjuvant therapy permitted)
* Prior STS therapy with ifosfamide or cyclophosphamide or other nitrogen mustards; prior systemic therapy with an anthracycline or anthracenedione; or prior mediastinal/cardiac radiotherapy
* Current use of drugs with known cardiotoxicity or known interactions with doxorubicin
* Anti-cancer treatment with radiation therapy, neoadjuvant or adjuvant chemotherapy, targeted therapies, immunotherapy, hormones or other antitumor therapies within 4 weeks prior to trial entry (6 weeks for nitrosoureas or mitomycin C).
* Significant cardiac dysfunction precluding treatment with doxorubicin as specified in the protocol
* Seizure disorders requiring anticonvulsant therapy unless seizure-free for the last year
* Known brain metastases (unless previously treated and well controlled for a period of >=3 months before screening)
* Previously diagnosed malignancies, except for adequately treated non-melanoma skin cancer, in situ cancer, or other cancer from which the subject has been disease-free for at least 5 years before screening
* Severe chronic obstructive or other pulmonary disease with hypoxemia (requires supplementary oxygen, symptoms due to hypoxemia or oxygen saturation <90% by pulse oximetry after a 2 minute walk) or in the opinion of the investigator any physiological state likely to cause normal tissue hypoxia
* Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1, without complete recovery
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Prior therapy with a hypoxic cytotoxin
* Subjects who participated in an investigational drug or device trial within 28 days prior to trial entry
* Known infection with human immunodeficiency virus (HIV) or active infection with hepatitis B or hepatitis C
* Subjects who have exhibited allergic reactions to a structural compound similar to TH-302 or the drug product excipients
* Subjects who are taking medications that prolong QT interval and have a risk of Torsades de Pointes
* Subjects with a corrected QT (QTc) interval calculated according to Bazett's formula of >450 milliseconds (msec) based on a screening electrocardiogram (ECG)
* Subjects with a history of long QT syndrome
* Subjects taking a medication that is a moderate or strong inhibitor or inducer of cytochrome P450 3A4 (CYP3A4)
* Females who are pregnant or breast-feeding
* Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
* Unwillingness or inability to comply with the study protocol for any reason
* Legal incapacity or limited legal capacity

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-12-10 (Actual); Primary Completion 2016-01-12 (Actual); Study Completion 2016-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono Co., Ltd., Japan
Locations (2):
- Japan (2):
  - Research Site, Kashiwa
  - Research Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/Last subject (informed consent): 10 December 2014/02 November 2015. Study completion date: 12 January 2016. Clinical data cut-off: 31 March 2016.
Pre-assignment Details: The study was planned to include a combination therapy period (including an initial Safety Run-In Phase followed by Phase II treatment period) and a TH-302 monotherapy period. However, due to early termination, only Safety Run-In Phase was conducted; thus, all the analyses are limited to Safety Run-In Phase.
Groups:
- TH-302 and Doxorubicin: Subjects received TH-302 at a dose of 300 milligram per square meter (mg/m^2) by intravenous infusion over 30 minutes on Day 1 and 8 of every 21-day cycle and Doxorubicin at a dose of 75 mg/m^2 by intravenous injection (over at least 5 minutes) or by intravenous infusion over 6-96 hours on Day 1 of every 21-day cycle starting 2 to 4 hours after completion of TH-302 administration until the evidence of significant treatment-related toxicity or progressive disease.
Period: Overall Study
Arm/Group | TH-302 and Doxorubicin
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF) included all subjects who received at least 1 dose of either TH-302 or doxorubicin.
Arm/Group | TH-302 and Doxorubicin
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (10.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) by Independent Central Review (Phase II Treatment Period)
Description: PFS was planned to assess as per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). Progressive Disease is defined as at least a 20 percent (%) increase in the Sum of longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: From first dose of study drug administration until PD or death, evaluated at 6 months
Population: As the study was terminated early following the discontinuation of the TH-302 clinical development program, it was decided as per Statistical Analysis Plan not to collect and evaluate the efficacy data for this study
Arm/Group | TH-302 and Doxorubicin
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression Free Survival (PFS) by Investigator Review (Phase II Treatment Period)
Description: PFS was planned to assess as per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). Progressive Disease (PD) is defined as at least a 20 percent (%) increase in the Sum of longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: From first dose of study drug administration until PD or death, evaluated at 6 months
Population: as for outcome 1
Arm/Group | TH-302 and Doxorubicin
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-free Survival (PFS) by Investigator and Independent Central Review (Phase II Treatment Period)
Description: as for outcome 2
Time Frame: From first dose of study drug administration until PD or death, evaluated at 3 months and 9 months
Population: as for outcome 1
Arm/Group | TH-302 and Doxorubicin
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-free Survival (PFS) (Phase II Treatment Period)
Description: as for outcome 2
Time Frame: From first dose of study drug administration until PD or death, assessed up to 12 months
Population: as for outcome 1
Arm/Group | TH-302 and Doxorubicin
Number analyzed (Participants) | 0

5. Secondary Outcome: Best Overall Response (BOR) by Independent Central Review (Phase II Treatment Period)
Description: BOR was planned to be determine according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) and as adjudicated by an Independent Central Review. BOR is defined as the best response of any of complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD) recorded from date of randomization until disease progression or recurrence (taking the smallest measurement recorded since start of treatment as reference). CR: Disappearance of all evidence of target and non-target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 millimeter (mm). PR: At least 30 percent (%) reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Stable disease (SD)=Neither sufficient increase to qualify for PD nor sufficient shrinkage to qualify for PR. PD is defined as at least a 20 % increase in the SLD, taking as reference the smallest SLD recorded from baseline or appearance of 1 or more new lesions.
Time Frame: From first dose of study drug administration until PD or death, assessed up to 12 months
Population: as for outcome 1
Arm/Group | TH-302 and Doxorubicin
Number analyzed (Participants) | 0

6. Secondary Outcome: Best Overall Response (BOR) by Investigator (Phase II Treatment Period)
Description: as for outcome 5
Time Frame: From first dose of study drug administration until PD or death, assessed up to 12 months
Population: as for outcome 1
Arm/Group | TH-302 and Doxorubicin
Number analyzed (Participants) | 0

7. Secondary Outcome: Duration of Response (Phase II Treatment Period)
Description: Duration of response according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) is defined as the time from the first assessment of complete response (CR) or partial response (PR) until the date of the first occurrence of progressive disease (PD), or until the date of death. CR: Disappearance of all evidence of target and non-target lesions. Any pathological lymph nodes must have reduction in short axis to less than (<) 10 millimeter (mm). PR: At least 30 percent (%) reduction from baseline in the sum of the longest diameter (SLD) of all lesions. PD is defined as at least a 20 percent (%) increase in the sum of the longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: From first dose of study drug administration until PD or death, assessed up to 12 months
Population: as for outcome 1
Arm/Group | TH-302 and Doxorubicin
Number analyzed (Participants) | 0

8. Secondary Outcome: Overall Survival (OS) (Phase II Treatment Period)
Description: OS is defined as the time from first dose to death due to any cause.
Time Frame: From first dose of study drug administration until the last subject completes the survival follow-up, assessed up to 12 months
Population: as for outcome 1
Arm/Group | TH-302 and Doxorubicin
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) (Safety Run-In Phase)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a subject which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. The term TEAE is defined as AEs starting or worsening after the first intake of the stud drug.
Time Frame: From baseline until end of trial, assessed up to Day 210
Population: The SAF Analysis Set included all subjects who received at least 1 dose of either TH-302 or doxorubicin.
Measure: Number; unit: Subjects
Arm/Group | TH-302 and Doxorubicin
Number analyzed (Participants) | 6
Subjects
  TEAEs | 6
  Serious TEAEs | 4

ADVERSE EVENTS:
Time Frame: Baseline up to Day 210 (Safety Run-In Phase)
Arm/Group | TH-302 and Doxorubicin
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TH-302 and Doxorubicin (N=6)
Pneumonia (Infections and infestations) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TH-302 and Doxorubicin (N=6)
Infection (Infections and infestations) | 1
Lymph gland infection (Infections and infestations) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Stomatitis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 4
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Fatigue (General disorders) | 2
Infusion site reaction (General disorders) | 1
Pyrexia (General disorders) | 4
Blood alkaline phosphatase increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 3
White blood cell count decreased (Investigations) | 3
Incorrect dosage administered (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1

LIMITATIONS AND CAVEATS:
This study was terminated early following the discontinuation of TH-302 clinical development program. Only 6 subjects were enrolled and treated in the Safety Run-In Phase; thus, the statistical analyses are limited to the Safety Run-In Phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other